CLINICAL TRIAL: NCT01522794
Title: Randomized Double Blind Placebo Controlled PK/PD Study on the Effects of a Single Intravenous Dose of NOX-H94 on Serum Iron During Experimental Human Endotoxemia
Brief Title: Pharmacokinetics/Pharmacodynamics of NOX-H94 in the Human Endotoxemia Model
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TME Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNOXH94C101; 2011-005022-22 (EudraCT Number)
Record Dates: First submitted 2012-01-18; First posted 2012-02-01 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Anemia of Chronic Disease
MeSH Terms: interventions — NOX-H94

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NOX-H94 (Experimental): Single dose of NOX-H94
  Interventions: Drug: NOX-H94
- Placebo (Placebo Comparator): Single dose of placebo control
  Interventions: Drug: Placebo solution

INTERVENTIONS:
Drug: NOX-H94 — single i.v. infusion
  Other Names: lexaptepid pegol
  Arms: NOX-H94
Drug: Placebo solution — single i.v. infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of the anti-hepcidin Spiegelmer NOX-H94 on iron homeostasis during systemic inflammation induced by endotoxin.

In the human endotoxemia model, intravenously administered lipopolysaccharide elicits an inflammatory response with release of pro-inflammatory cytokines, such as IL-6 and TNF-alfa, with subsequent induction of hepcidin. As a consequence of hepcidin induction, serum iron concentrations decrease.

This study in healthy subjects investigates the capacity of NOX-H94 to inactivate hepcidin and to prevent serum iron decrease in a pathophysiological model prior to studying the efficacy of NOX-H94 in patients with anemia of chronic disease.

ELIGIBILITY:
Main Inclusion Criteria:

* BMI between 18 and 30 kg/m², with a lower limit of body weight of 50 kg
* Healthy as determined by medical history, physical examination, vital signs, 12 lead electrocardiogram, and clinical laboratory parameters
* Serum iron and red blood parameters Hb, MCV, ferritin, serum iron, and total iron binding capacity within reference range

Main Exclusion Criteria:

* Use of any medication, recreational drugs or anti-oxidant vitamin supplements within 7 days
* Use of caffeine, nicotine, or alcohol within 1 day
* Previous participation in a trial where LPS was administered
* Surgery or trauma with significant blood loss or blood donation within 3 months
* History, signs or symptoms of cardiovascular disease (vaso-vagal collapse or of orthostatic hypotension, Resting pulse rate ≤45 or ≥100/min, Hypertension, Hypotension, ECG conduction abnormalities)
* Renal impairment: plasma creatinine >120 µmol/L
* Liver function tests (alkaline phosphatase, AST, ALT and γ-GT) outside of the reference range or total bilirubin >20 µmol/L
* Hemoglobin or iron parameters (iron, transferring saturation, ferritin) outside of the reference ranges
* History of asthma
* Immuno-deficiency
* Positive test of HIV type 1/2 antibodies, HBs antigen, HBc antibodies and HCV antibodies unless antibody titer is induced by vaccination
* CRP > reference range or clinically significant acute illness, including infections, within 2 weeks
* Treatment with investigational drugs or participation in any other clinical trial within 30 days prior to study drug administration
* Known or suspected of not being able to comply with the trial protocol
* Inability to personally provide written informed consent and/or take part in the study

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
serum iron | 9 hours
  Change versus baseline; comparison of subjects treated with NOX-H94 versus placebo

SECONDARY OUTCOMES:
Pharmacodynamics: Effects of NOX-H94 on Iron homeostasis | up to 2 Weeks
  Change from baseline and group comparison (NOX-H94 vs. placebo) of:
  serum iron, transferrin saturation, ferritin
Pharmacokinetic profile of NOX-H94 | 12 time points over 2 Weeks
  plasma concentration-time profile T0 to 2 weeks
Safety and tolerability | up to 2 Weeks
  Safety and tolerability parameters will be evaluated along the entire study duration consisting of spontaneously reported adverse events, physical examination and vital signs, hematology and clinical chemistry laboratory examinations.
Effects of NOX-H94 on innate immune response | up to 2 weeks
  To assess the effect of a single dose administration of NOX H94 on the innate immune response during experimental endotoxemia: TNF-α, IL-6, IL-1RA, IL-10
Pharmacokinetics: Cmax of NOX-H94 | Day 1
Pharmacokinetics: AUC of NOX-H94 | 0-2 weeks
Pharmacokinetics: Clearance of NOX-H94 | 0-2 weeks
Pharmacodynamics: effect of NOX-H94 on Red blood cell parameters | 0- 2 weeks
  Change versus baseline and group comparison: reticulocyte hemoglobin content, hemoglobin, mean cell volume, mean cell hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Kai Riecke, MD, Study Director — TME Pharma AG; Peter Pickkers, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] van Eijk LT, John AS, Schwoebel F, Summo L, Vauleon S, Zollner S, Laarakkers CM, Kox M, van der Hoeven JG, Swinkels DW, Riecke K, Pickkers P. Effect of the antihepcidin Spiegelmer lexaptepid on inflammation-induced decrease in serum iron in humans. Blood. 2014 Oct 23;124(17):2643-6. doi: 10.1182/blood-2014-03-559484. Epub 2014 Aug 27. PMID 25163699
- See also: Result summary: Abstract 3452, ASH 2012 — https://ash.confex.com/ash/2012/webprogram/Paper50672.html